CLINICAL TRIAL: NCT02735577
Title: Neurocognitive Mechanisms of Disulfiram Treatment of Alcohol Use Disorder
Brief Title: Neural Mechanisms of Disulfiram Effects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Nasir Naqvi, research psychiatrist, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 7193
Record Dates: First submitted 2016-04-06; First posted 2016-04-12 (Estimated); Results first posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-10

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol; Craving; Functional MRI; Cognitive control; Risky decision-making; Disulfiram
MeSH Terms: conditions — Alcoholism | interventions — Disulfiram

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Disulfiram (Experimental): Patients in this arm will receive disulfiram 250 mg daily for a total of 40 days.
  Interventions: Drug: Disulfiram

INTERVENTIONS:
Drug: Disulfiram — Patients will be hospitalized on an inpatient psychiatric unit for 1-7 days to initiate abstinence. An fMRI scan will be performed to examine neural mechanisms of alcohol motivation. Prior to discharge, patients will receive the first dose of disulfiram 500 mg. They will then attend an outpatient clinic every other day for 14 days. At each clinic visit, they will receive 500 mg of disulfiram under supervision. Another fMRI scan examining alcohol motivation will be performed. Following this, all patients will attend the clinic weekly, and will be prescribed disulfiram 250 mg daily to take at home. This will be followed followed by an optional extension of weekly visits taking disulfiram 250 mg daily for another 28 days, for a total of 70 days of disulfiram treatment.
  Other Names: Antabuse

SUMMARY:
This study combines functional MRI with medication treatment in order to understand the neural mechanisms by which disulfiram, a currently approved medication for alcohol use disorder, changes behavior. Disulfiram is a medication that prevents drinking by causing a highly unpleasant physical reaction when alcohol is consumed while it is being taken. Thus, it provides a means for studying the general neural mechanisms by which awareness of risks impacts behavior change in alcohol use disorder.

DETAILED DESCRIPTION:
The overall goal of this project is to combine functional brain imaging and clinical methods in order to examine how treatment with disulfiram (DIS) alters neural activity related to alcohol-seeking motivation in patients with alcohol use disorder (AUD). DIS is an established, effective, FDA-approved medication for AUD that causes a highly aversive physical reaction if alcohol is consumed while it is being taken. The mere awareness of the risk or threat the DIS-alcohol reaction deters alcohol use, i.e. it is not necessary to drink alcohol while taking DIS to change behavior. By uncovering the neural mechanisms underlying this risk/threat-based psychological effect, it will be possible to integrate DIS with biologically based treatments targeted at these neural mechanisms, with the goal of improving the efficacy of DIS. Furthermore, the results will shed light on the general neural mechanisms by which awareness of risks of substance use impacts addictive motivation. This is a core process in a number of behavioral treatments for substance use disorders, such as Motivational Interviewing and Contingency Management, as well as in behavior change in non-treatment settings.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 21-60
2. Right-handed
3. Capable of giving informed consent and complying with study procedures
4. Reports drinking a minimum of 5 standard drinks for men or 4 standard drinks for women on at least 4 days per week on average over the past 28 days
5. Meets DSM-V criteria for current Alcohol Use Disorder
6. Seeking treatment for Alcohol Use Disorder
7. Agree to not seek additional treatment, apart from Alcoholics Anonymous
8. Willing to attempt to abstain from alcohol completely for the duration of the study
9. Willing to be hospitalized on a research unit for 24 hours, longer if detoxification is needed.

Exclusion Criteria:

1. Risk of severe alcohol withdrawal (e.g. history of seizures or delirium tremens)
2. Current Moderate or Severe Substance Use Disorder, other than Alcohol, Nicotine or Caffeine Use Disorders
3. Lifetime history of Bipolar Disorder, Schizophrenia or Schizoaffective Disorder
4. Any current psychiatric disorder, other than Alcohol Use Disorder, that, in the judgment of the investigator, will require treatment that will interfere with study participation.
5. Current severe depression (HAM-D >24) or anxiety (HAM-A >24)
6. Significant suicide or violence risk
7. Currently taking any psychotropic medications
8. Legally mandated to participate in treatment
9. History of prior treatment with disulfiram
10. Sufficiently socially unstable as to preclude participation (e.g. homeless)
11. Contraindications to disulfiram treatment (liver disease, kidney disease, cardiac disease, seizure disorder, hypothyroidism, diabetes mellitus, pregnancy or lactation, allergy to disulfiram or thiuran derivatives)
12. Neurological or medical conditions that would interfere with MRI scanning (e.g. history of stroke, seizure, brain tumor, brain infection, traumatic brain injury, multiple sclerosis, dementia, metal device in body, pregnancy, claustrophobia, color blindness, severe hearing impairment, weight>300 lbs., wheelchair-bound)
13. Currently taking medications containing alcohol, metronidazole, isoniazid, paraldehyde, phenytoin, warfarin, or theophylline.
14. Significant alcohol withdrawal (CIWA>8) at screening, after confirming a blood alcohol level of zero.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2016-03; Primary Completion 2019-10-31 (Actual); Study Completion 2020-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nasir H. Naqvi, MD, PhD, Principal Investigator — NYP Institute
Locations (1):
- NYPInstitute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saifi MA, Shaikh AS, Kaki VR, Godugu C. Disulfiram prevents collagen crosslinking and inhibits renal fibrosis by inhibiting lysyl oxidase enzymes. J Cell Physiol. 2022 May;237(5):2516-2527. doi: 10.1002/jcp.30717. Epub 2022 Mar 13. PMID 35285015

RESULTS

PARTICIPANT FLOW:
Groups:
- Disulfiram: Patients in this arm will receive disulfiram 250 mg daily for a total of 42 days.
  Disulfiram: Patients will be hospitalized on an inpatient psychiatric unit for 1-7 days to initiate abstinence. An fMRI scan will be performed to examine neural mechanisms of alcohol motivation. Prior to discharge, patients will receive the first dose of disulfiram 500 mg. They will then attend an outpatient clinic every other day for 14 days. At each clinic visit, they will receive 500 mg of disulfiram under supervision. Another fMRI scan examining alcohol motivation will be performed. Following this, all patients will attend the clinic weekly, and will be prescribed disulfiram 250 mg daily to take at home. This will be followed followed by an optional extension of weekly visits taking disulfiram 250 mg daily for another 28 days, for a total of 70 days of disulfiram treatment.
Period: Disulfiram Treatment
Arm/Group | Disulfiram
Started | 7
Completed | 6
Not Completed | 1
Not completed — Lost to Follow-up | 1
Period: Optional 28 Days of Disulfiram Treatment
Arm/Group | Disulfiram
Started | 6
Completed | 4
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Enrolled Participants
Arm/Group | Disulfiram
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 2
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 7
Baseline Drinking days (prior 28 days) [Mean (Standard Deviation); unit: days] | 24.0 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Use
Description: Number of drinking days
Time Frame: 42 days
Population: Participants who completed the initial 42 days of disulfiram treatment
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Disulfiram
Number analyzed (Participants) | 6
days | 0 (0)

ADVERSE EVENTS:
Time Frame: 42 days of initial disulfiram treatment or length of participation
Arm/Group | Disulfiram
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

LIMITATIONS AND CAVEATS:
fMRI data analysis is not complete because there are not enough subjects to produce valid data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-01-26): https://cdn.clinicaltrials.gov/large-docs/77/NCT02735577/Prot_000.pdf
  • Statistical Analysis Plan (2014-11-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT02735577/SAP_001.pdf